CLINICAL TRIAL: NCT00214097
Title: Phase I/II Trial Examining Dose-per-Fraction Escalation Using Intensity Modulated Radiation Therapy in the Treatment of Prostate Cancer
Brief Title: Phase I/II Hypofractionated Radiotherapy for Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RO02803; NCI (P01 CA88960); 2002-322 (Other: Institutional Review Board); A533300 (Other: UW Madison); SMPH/HUMAN ONCOLOGY (Other: UW Madison)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: dose escalation, 3 possible dose groups, with one Phase II group based on MTD.
  Per protocol, while waiting for safety data to mature for escalation, protocol permitted enrollment to continue on last dose that was already proven safe. Thus Arms one and two have more than 50 subjects each.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Level 1 (Experimental): 64.7 Gy/22 fractions of 2.94 Gy
  Interventions: Radiation: Radiotherapy
- Level 2 (Experimental): 58.08 Gy/16 fractions of 3.63 Gy
  Interventions: Radiation: Radiotherapy
- Level 3 (Experimental): 51.6 Gy/12 fractions of 4.3 Gy
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Daily radiation to prescribed dose

SUMMARY:
The purpose of this study is to examine the clinical feasibility of using Intensity-modulated radiation therapy (IMRT) combined with daily pretreatment prostate localization to deliver increasingly hypofractionated treatment courses. Progressively larger fraction sizes will be delivered in a phase I design based on both acute and long-term tolerances to the treatment. The dose-per-fraction escalation design utilizes schemas that maintain an isoeffective dose for late effects, while predicting that tumor control will actually improve. The delivery of fewer, larger fractions of radiation, if proven effective and safe, would result in significant cost saving and more efficient use of resources. Phase II will commence with Maximum Tolerated Dose (MTD) finding with up to 200 additional patients being enrolled during this phase of the study.

ELIGIBILITY:
Inclusion Criteria:

Histologically proven adenocarcinoma of the prostate.

* Stage ≤ T2b disease, as defined by 1997 American Joint Committee on Cancer (AJCC) classification
* Predicted risk of lymph node involvement (by standard nomograms) of 15% or less (24), OR histologically negative pelvic nodes
* Gleason score ≤ 7
* No evidence of distant metastasis
* Age 18+
* Informed consent signed in accordance with institutional protocol
* Pretreatment evaluations must be completed as specified in Section 7.0.
* ECOG performance status 0-1
* No previous or concurrent cancers, other than localized basal cell or squamous cell skin carcinoma, unless continually disease free for at least 5 years
* No prior pelvic irradiation, prostate brachytherapy, or bilateral orchiectomy
* Gonadotropin-releasing hormone agonist (GnRH-a) use permitted (maximum of 6 months duration). Anti-androgen therapy permitted concurrently with GnRH-a.
* No previous or concurrent cytotoxic chemotherapy
* No radical surgery or cryosurgery for prostate cancer
* The absence of any co-morbid medical condition which would constitute a contraindication for radical radiotherapy
* The absence of serious concurrent illness of psychological, familial, sociological, geographical or other concomitant conditions which do not permit adequate follow-up and compliance with the study protocol.
* No current use of anticoagulation therapy, other than aspirin.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2002-10-14 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2017-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ritter, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Result] Brower JV, Forman JD, Kupelian PA, Petereit DG, Gondi V, Lawton CA, Anger N, Saha S, Chappell R, Ritter MA. Quality of life outcomes from a dose-per-fraction escalation trial of hypofractionation in prostate cancer. Radiother Oncol. 2016 Jan;118(1):99-104. doi: 10.1016/j.radonc.2015.12.018. Epub 2016 Jan 2. PMID 26755165
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Level 1: 2.94 gy/fr, 22 fractions,
  Radiotherapy: Daily radiation to prescribed dose
- Level 2: 3.63 gy/fr, 16 fractions, 50 patients first 10 treated with 4 fractions per week next 40 treated with 5 fractions per week
  Radiotherapy: Daily radiation to prescribed dose
- Level 3: 4.3 gy/fr, 12 fractions, 50 patients first 10 treated with 4 fractions per week next 40 treated with 5 fractions per week
  Radiotherapy: Daily radiation to prescribed dose
Period: Overall Study
Arm/Group | Level 1 | Level 2 | Level 3
Started | 101 (Escalation to the next higher level will occur when > 20 pt yrs of F/U and > 5 pts followed >1 yr) | 111 (Escalation to the next higher level will occur when > 20 pt yrs of F/U and > 5 pts followed >1 yr) | 135
Completed | 101 | 111 | 135
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Level I: 2.94 gy/fr, 22 fractions,
  Radiotherapy: Daily radiation to prescribed dose
- Level II: 3.63 gy/fr, 16 fractions,
  Radiotherapy: Daily radiation to prescribed dose
- Level III: 4.3 gy/fr, 12 fractions,
  Radiotherapy: Daily radiation to prescribed dose
- Total: Total of all reporting groups
Arm/Group | Level I | Level II | Level III | Total
Number analyzed (Participants) | 101 | 111 | 135 | 347
Age, Continuous [Median (Full Range); unit: years] | 67 [47 to 83] | 67 [45 to 81] | 68 [52 to 85] | 68 [45 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 101 | 111 | 135 | 347
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 76 | 98 | 118 | 292
  Unknown or Not Reported | 25 | 11 | 15 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 78 | 84 | 108 | 270
  Black | 5 | 16 | 10 | 31
  Unknown | 17 | 11 | 17 | 45
  Asian | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 101 | 111 | 135 | 347

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience Grade 3 or Higher Acute Toxicities
Description: To evaluate acute tolerances to dose-per-fraction escalation in the treatment of prostate cancer using optimized treatment of Intensity-modulated radiation therapy (IMRT), daily rectal balloon displacement, and transabdominal ultrasound localization of the prostate. For toxicities observed within the first 10 patients at each hypofractionation level, ≥20% acute grade 3 or higher GI or genitourinary (GU) toxicity will constitute a threshold toxicity level and will dictate a decrease in frequency of treatment by one treatment per week. Maximum tolerated dose is reached if 20% of participants experience acute toxicities grade 3 or higher.
Time Frame: 90 days post radiation treatment
Measure: Count of Participants; unit: Participants
Groups:
- Level 2: 3.63 gy/fr, 16 fractions,
  Radiotherapy: Daily radiation to prescribed dose
- Level 3: 4.3 gy/fr, 12 fractions,
  Radiotherapy: Daily radiation to prescribed dose
Arm/Group | Level 1 | Level 2 | Level 3
Number analyzed (Participants) | 101 | 111 | 135
Participants | 1 | 1 | 0

2. Primary Outcome: Number of Subjects Experiencing Grade 2 or Higher Late Rectal Toxicities at Any Time During Follow Up
Description: To evaluate late radiation toxicities to dose-per fraction escalation in the treatment of prostate
Time Frame: from 90 days post XRT through last follow-up visit (up to 3 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Level I | Level II | Level III
Number analyzed (Participants) | 101 | 111 | 135
Participants | 14 | 26 | 29

3. Secondary Outcome: Biochemical Progression-free Survival Based on PSA Surveillance
Description: Patients will be considered to be without biochemical recurrence if either the Prostate-specific antigen (PSA) is still declining or the PSA nadir has been reached and is below 1.0ng/ml
Time Frame: up to 15 years from enrollment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Level I | Level II | Level III
Number analyzed (Participants) | 101 | 111 | 135
percentage of participants | 91.5 [88.2 to 94.8] | 92.7 [90 to 95.4] | 94.1 [91.9 to 96.3]

4. Secondary Outcome: Fox Chase Bowel Survey at Baseline and 3 Years
Description: The Fox Chase Bowel/Bladder survey was divided into two sections: Bowel (questions 1 to 14, N=14) and Bladder (questions 19, and 21 to 30, N=11). To facilitate analysis, Bowel and Bladder scores for each section were rescaled to a total score of between 0 - 100, where higher scores indicated better Quality of Life (QoL). Results for the Bowel Section are reported here.
Time Frame: Baseline and 3 years
Population: Unavailable quality of life questionnaires at year 3. All mean scores were adjusted for missing data. The missing data for questionnaires were handled by weighted mean imputation. Cases with more than half of the total questions missing were not included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Level I: 2.94 gy/fr, 22 fractions
  Radiotherapy: Daily radiation to prescribed dose
- Level II: 3.63 gy/fr, 16 fractions
  Radiotherapy: Daily radiation to prescribed dose
- Level III: 4.3 gy/fr, 12 fractions
  Radiotherapy: Daily radiation to prescribed dose
Arm/Group | Level I | Level II | Level III
Number analyzed (Participants) | 101 | 111 | 135
scores on a scale
  Baseline | 90.0 (10.7) | 88.0 (14.6) | 86.2 (14.6)
  Year 3: number analyzed (Participants) | 45 | 48 | 57
  Year 3 | 86.3 (11.1) | 87.7 (11.6) | 85.4 (14.7)

5. Secondary Outcome: Fox Chase Bladder Survey at Baseline and 3 Years
Description: The Fox Chase Bowel/Bladder survey was divided into two sections: Bowel (questions 1 to 14, N=14) and Bladder (questions 19, and 21 to 30, N=11). To facilitate analysis, Bowel and Bladder scores for each section were rescaled to a total score of between 0 - 100, where higher scores indicated better Quality of Life. Results for the Bladder Section are reported here.
Time Frame: Baseline and 3 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Level I | Level II | Level III
Number analyzed (Participants) | 101 | 111 | 135
scores on a scale
  Baseline | 84.2 (9.4) | 84.7 (10.1) | 82.7 (11.3)
  3 years: number analyzed (Participants) | 45 | 48 | 57
  3 years | 79.5 (13.5) | 82.5 (10.1) | 81.1 (12.2)

6. Secondary Outcome: International Index of Erectile Function (IIEF) Score at Baseline and 3 Years
Description: The IIEF is a 15-item survey where 9-items are scored 0-5 and 6-items are scored 1-5 with a total range of 6-75. The standard scoring mechanism was used for IIEF, where the QoL items corresponded to the following domains: erectile function (score range 1-30), orgasmic function (score range 1-10), sexual desire (score range 2-10), intercourse satisfaction (score range 0-15), and overall satisfaction (score range 2-10). Higher numbers indicate increased QoL.
Time Frame: Baseline and 3 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Level I | Level II | Level III
Number analyzed (Participants) | 101 | 111 | 135
scores on a scale
  Baseline | 15.6 (11.7) | 17.6 (11.7) | 15.1 (11.1)
  3 years: number analyzed (Participants) | 41 | 43 | 51
  3 years | 10.4 (10.6) | 13.6 (11.7) | 9.6 (8.9)

7. Secondary Outcome: Spritzer Quality of Life Index (SQLI) at Baseline and 3 Years
Description: The SQLI is composed of five items (activity, daily living, health, support, outlook) scored utilizing a numerical scale of 0-2. Standard scoring was also used for the SQLI survey (total score range 0-10) where higher score indicate increased QoL.
Time Frame: Baseline and 3 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Level I | Level II | Level III
Number analyzed (Participants) | 101 | 111 | 135
scores on a scale
  Baseline | 9.7 (0.7) | 9.4 (1.2) | 9.5 (1.4)
  Year 3: number analyzed (Participants) | 44 | 47 | 55
  Year 3 | 9.5 (1.4) | 9.8 (0.4) | 9.5 (1.4)

ADVERSE EVENTS:
Time Frame: Acute GI and GU toxicities and Late GI and GU toxicities were recorded for the duration of the study. For level 1 patients, median followup was 100 months, for level 2 patients median follow up was 85.5 months and for level 3 it was 61.7 months
Groups:
- Level 1: 2.94 gy/fr, 22 fractions, minimum 50 patients to escalate, (back filling permitted while next dose level data matures for escalation) first 10 treated with 4 fractions per week next 40 + treated with 5 fractions per week
  Radiotherapy: Daily radiation to prescribed dose
- Level 2: 3.63 gy/fr, 16 fractions, minimum 50 patients ( back filling permitted while next dose level data matures for escalation) first 10 treated with 4 fractions per week next 40 + treated with 5 fractions per week
  Radiotherapy: Daily radiation to prescribed dose
- Level 3: 4.3 gy/fr, 12 fractions, 50 patients, for safety, up to an additional 100 for phase II component of study first 10 treated with 4 fractions per week next 40 +treated with 5 fractions per week
  Radiotherapy: Daily radiation to prescribed dose
Arm/Group | Level 1 | Level 2 | Level 3
All-Cause Mortality (participants affected / at risk) | 22/101 | 18/111 | 20/135
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/111 | 0/135
Other Adverse Events (participants affected / at risk) | 40/101 | 56/111 | 52/135
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level 1 (N=101) | Level 2 (N=111) | Level 3 (N=135)
Acute GI (Gastrointestinal disorders) | 3 (3) | 6 (6) | 3 (3) — modified RTOG grading criteria
Acute GU (Renal and urinary disorders) | 23 (23) | 24 (24) | 20 (20) — RTOG modified grading criteria
Late GI and GU toxicities (Renal and urinary disorders) | 14 (14) | 26 (26) | 29 (29) — FC-LENT grading criteria

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2006-01-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT00214097/Prot_SAP_000.pdf